CLINICAL TRIAL: NCT01950260
Title: Prevention of Overt Hypothyroidism Following Radioactive Iodine Therapy for Graves' Disease
Brief Title: Early Levothyroxine Post Radioactive Iodine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marius Stan, Associate Professor of Medicine, Endocrinology Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13-002570
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Graves' Disease
Keywords: Graves' disease; Radioactive iodine; Hypothyroidism
MeSH Terms: conditions — Graves Disease; Hypothyroidism | interventions — Thyroxine; Thyroid Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxine (Experimental): In the intervention arm patients will start levothyroxine therapy at 4 weeks after RAI therapy. The initial dose of levothyroxine will be 25 mcg/day. It will be increased to 50 mcg/day 2 weeks later and then adjusted at 8 weeks post RAI based on a full face-to-face clinical and biochemical evaluation.
  Interventions: Drug: Levothyroxine
- Placebo (Placebo Comparator): In the control arm patients will receive placebo capsules and be evaluated for levothyroxine therapy during a full face-to-face evaluation at 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levothyroxine — Early initiation of levothyroxine after radioactive iodine (to start at 4 weeks).
  Other Names: Thyroid hormone
  Arms: Levothyroxine
Other: Placebo — Placebo to start at 4 weeks after RAI
  Arms: Placebo

SUMMARY:
The study will try to answer the question of whether early treatment with levothyroxine at 4 weeks after radioactive iodine for Graves'disease will prevent overt hypothyroidism (low thyroid hormone levels).

ELIGIBILITY:
Inclusion criteria:

-all adult patients (ages 18-70 years) with Graves' Disease (GD) who will receive radioactive iodine (RAI) ablation of the thyroid gland for treatment of GD

Exclusion criteria:

* clinically manifest Graves' ophthalmopathy (GO)
* recent (<1 yr.) history of arrhythmias or any history of ventricular arrhythmias
* preexistent cardiomyopathy
* malnutrition
* psychiatric history that could get worse if patient remains persistently hyperthyroid
* unlikely to return for the planned follow-up visits
* unlikely to comply with the blood drawing schedule
* unlikely to complete the hypothyroid-Health Related Quality of Life (HDQL) and Thyroid Specific (TSQ) questionnaires

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Stan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Levothyroxine | Placebo
Started | 30 | 31
Completed | 30 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levothyroxine | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (15) | 48 (13) | 47.5 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61
Weight [Mean (Standard Deviation); unit: kg] | 68.5 (16.6) | 73.4 (17.5) | 70.9 (17)
Thyroid size [Mean (Standard Deviation); unit: grams] | 32.7 (10.8) | 31.4 (13.9) | 32 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overt Hypothyroidism
Description: Incidence of overt hypothyroidism at 8 weeks post radioactive iodine treatment (RAI). Overt hypothyroidism was defined as thyroid stimulating hormone (TSH) test result > 3.0 milliunits per liter (mIU/L) or thyroid hormone free T4 (fT4) < 0.8 nanograms per deciliter (ng/dL). Free T4 is the portion of total T4 thyroid hormone that is available to your tissues in your bloodstream.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Levothyroxine | Placebo
Number analyzed (Participants) | 30 | 31
Participants | 11 | 17
Statistical Analysis 1: Comparison: Levothyroxine vs Placebo; Test type: Superiority; p = 0.23, Fisher Exact

2. Secondary Outcome: Change in Hypothyroid-Health Related Quality of Life
Description: The mean change in Quality of life scores was measured by the Hypothyroid-Health Related Quality of Life (HRQL) questionnaire. This questionnaire consists of 27 questions specifying the severity of the discomfort or symptoms of hypothyroidism using a 5 point scale for each question with "not at all"=1 to "all the time"=5. Higher scores are associated with a lower quality of life. The change between weeks 4 and 8 were assessed using a hierarchical linear model. The primary parameter of interest from the model was the treatment by time interaction term. Time was a collection of indicator values representing each assessment point.
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levothyroxine | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale | 12 (28.4) | 19.8 (25.0)
Statistical Analysis 1: Comparison: Levothyroxine vs Placebo; Test type: Superiority; p = 0.41, Regression, Linear

3. Secondary Outcome: Change in Thyroid Specific Quality of Life
Description: The mean change in quality of life scores was measured by the Thyroid Specific Questionnaire (TSQ). This questionnaire consists of 12 questions ranked on a four-point scale for each question where 0 is 'better than usual' and 3 is 'much less than usual'. A higher score indicates higher levels of dissatisfaction and a lower quality of life. The change between weeks 4 and 8 were assessed using a hierarchical linear model. The primary parameter of interest from the model was the treatment by time interaction term. Time was a collection of indicator values representing each assessment point.
Time Frame: 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Levothyroxine | Placebo
Number analyzed (Participants) | 30 | 31
units on a scale | -2 (12.8) | -3.8 (8.7)
Statistical Analysis 1: Comparison: Levothyroxine vs Placebo; Test type: Superiority; p = 0.33, Regression, Linear

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from enrollment until study completion, approximately 6 months.
Arm/Group | Levothyroxine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/31
Other Adverse Events (participants affected / at risk) | 3/30 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine (N=30) | Placebo (N=31)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levothyroxine (N=30) | Placebo (N=31)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT01950260/Prot_SAP_000.pdf